CLINICAL TRIAL: NCT01373970
Title: The Clinical Significance of Acid Rebound: Symptoms of Reflux After PPI Treatment in Patients With Functional Dyspepsia
Brief Title: The Clinical Significance of Acid Rebound in Functional Dyspepsia
Acronym: CLARIFY
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Anders Bergh Loedrup, Doctor, Zealand University Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SJ-217
Record Dates: First submitted 2011-05-17; First posted 2011-06-15 (Estimated); Last update posted 2013-12-06 (Estimated); Status verified 2013-12

CONDITIONS: Functional Dyspepsia
Keywords: Functional Dyspepsia; Protonpump inhibitor; Rebound Acid HyperSecretion
MeSH Terms: interventions — Pantoprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- PPI + Placebo (Active Comparator): PPI followed by cross over to placebo
  Interventions: Drug: Pantoprazole + Placebo

INTERVENTIONS:
Drug: Placebo — Placebo, one tablet daily for 12 weeks
  Arms: Placebo
Drug: Pantoprazole + Placebo — Pantoprazole 40 mg, one tablet daily in eight weeks followed by a blinded cross over to placebo, one tablet daily for four weeks
  Arms: PPI + Placebo

SUMMARY:
Proton pump inhibitors (PPI) have been shown to cause acid reflux related symptoms at withdrawal in healthy volunteers, a phenomenon known as Rebound Acid Hyper Secretion. Whether this also applies for patients with dyspeptic symptoms but without true reflux disease (functional dyspepsia) treated with PPI is unknown. If this is the case, it could lead to an unfortunate long term use of PPI, since the acid rebound renders withdrawal too difficult.

This is a single centre, randomized, double-blinded, placebo-controlled cross over study. Study period is 12 weeks per study subject. Study subjects are referred to the study from General Practitioner (GP) and the gastroenterology department or endoscopy clinic of the investigational centre.

The study population consists of patients who seek their GP because of dyspepsia without alert signs, and whom the GP may consider starting on PPI. Out patients referred to the gastroenterology department or endoscopy clinic of the investigational centre because of dyspepsia without specific exclusion criteria are also invited to participate.

Baseline interview, upper endoscopy and pH monitoring are performed one week before inclusion to exclude patients with GERD. Helicobacter Pylori (Hp.) status is assessed by Helicobacter Urease Test (HUT). Hp. positive subjects without ulcus are not excluded.

Patients with a positive pH monitoring will not be included in the analysis regarding the primary endpoint (Development of GERD) but will be included in the analysis regarding one of the secondary endpoints (Effect of PPI on Functional Dyspepsia).

Study subjects are randomized to either pantoprazol followed by cross over to placebo or to placebo. Escape medication in the form of Gaviscon can be used on demand.

Internet based questionnaires are answered weekly. Questionnaires consist of the Gastrointestinal Symptom rating Scale (GSRS) in combination with items assessing postprandial fullness and items assessing the Montreal Criteria for Gastro Esophageal Reflux Disease (GERD).

Compliance to protocol is assessed at hospital visits every fourth week. At the end of study endoscopy and pH monitoring are repeated.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms indicating dyspepsia, including:

  * Epigastric pain or epigastric discomfort
  * Bothersome postprandial fullness
  * Early satiation
  * Epigastric burning
* Access to internet

Exclusion Criteria:

* Daily use of PPI or H2-receptor antagonists in more than 28 days within the last 120 days OR more than two days within the last 28 days OR more than five non-consecutive days within the last 28 days.
* Mild heartburn or regurgitation more than once per week
* Moderate or severe heartburn or regurgitation at least once per week
* Complications to GERD (esophagitis, stricture or Barrett's esophagus) prior to enrolment or at screening
* Abnormal findings at upper endoscopy necessitating treatment
* Abnormal pH-monitoring prior to enrolment or at screening (pH <4 in ≥5.5 % of the time on "worst day" of 48-h monitoring)

  * Excludes data from analysis regarding primary endpoint (see summary)
* Previous surgery on esophagus, stomach or duodenum
* Regular use of NSAIDs through the last six months
* Potential language problems in understanding information and registering symptoms
* Pregnancy or breast feeding
* Other diseases which can interfere with the symptom registration (severe congestive heart disease, malignant disease, schizophrenia ect.)
* Abuse of alcohol/narcotics
* Allergy/intolerance to gelatine or lactose used in placebo
* Patients with pacemaker, Implantable Cardioverter Defibrillator or Implantable Neurostimulator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2011-05; Primary Completion 2013-05 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Development of GERD | week 9 - 12
  Comparison of number of study subjects that develop GERD according to the Montreal definition including endoscopic findings and pH monitoring in weeks 9-12 in the PPI group versus the placebo group.

SECONDARY OUTCOMES:
Use of escape medication | Week 9 - 12
  Difference in use of escape medication in weeks 9 - 12 between PPI- and placebo group
Endoscopic findings | 0 - 2 weeks before inclusion
  Number of study subjects who have esophagitis, peptic stricture or Barrett's esophagus at inclusion without having symptoms of reflux.
pH monitoring | 0 - 2 weeks before inclusion
  Number of study subject who have an abnormal pH monitoring at inclusion with-out symptoms of reflux
Irritable Bowel Syndrome (IBS) | 0 - 2 weeks before inclusion
  Number of study subjects with ROME III score indicating IBS at inclusion
Irritable Bowel Syndrome (IBS) and treatment | Week 0 - 12
  Difference in symptom scores between study subjects with and without IBS in the PPI- and placebo group in weeks 0 - 12
Effect of PPI on Functional Dyspepsia | Week 8
  Number of study subjects in the PPI group versus the placebo group that answer "no discomfort at all" or "slight discomfort" to dyspepsia related questions ("ache/pain in the upper part of the abdomen" and "hunger pains/hollow feeling in the stomach") in week 8.
Helicobacter Pylori | Week 9 - 12
  Difference in symptom score for subject with and without H. Pylori between PPI- and placebo group in weeks 9 - 12.

CONTACTS AND LOCATIONS:
Overall Officials: Anders B. Lødrup, MD, Principal Investigator — Zealand University Hospital
Locations (1):
- Koege Hospital, Koege, Denmark